CLINICAL TRIAL: NCT06195904
Title: Genomic Profiling of Pancreatic Cystic Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JooKyung Park, Associate professor, Samsung Medical Center
Other Study IDs: 2022-10-056; KC22TISI0829
Record Dates: First submitted 2023-11-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Pancreatic Cyst
MeSH Terms: conditions — Pancreatic Cyst | interventions — Sodium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Pancreatic cyst fluid Pancreatic cyst tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NA (No intervention) — NA (No intervention)

SUMMARY:
This study aims to find out whether quantitative and qualitative analysis, including genetic mutation analysis, of samples obtained from patients with pancreatic cysts is associated with the risk of malignancy, and helpful in the differential diagnosis of mucinous and serous cysts. The study design is a single-arm prospective cohort observational study. Using blood, pancreatic cyst fluid, and pancreatic cyst tissue, genetic mutation analysis and measurement of various biomarkers are performed, and the relationship between these and malignancy or whether they are helpful in distinguishing mucinous and serous cysts is analyzed. The primary outcome is genetic variants of pancreatic cysts associated with malignancy. The secondary outcomes are factors including genetic variants that differentiate mucinous from serous cysts.

DETAILED DESCRIPTION:
Pancreatic cysts, especially mucinous cysts, are precancerous lesions that can cause pancreatic cancer, and follow-up surveillance is important. However, there is a lack of clear medical evidence for the proper method and timing of follow-up, so the current follow-up strategies rely heavily on the opinions of experts. Although mucinous pancreatic cyst is known as a precancerous lesion, the incidence of cancer is about 1-5%. Therefore, if the risk of malignant disease can be more accurately predicted in patients with pancreatic cysts, patients with a high risk of malignant disease can be more intensively monitored and improved survival rates can be expected through early detection of pancreatic cancer. In addition, unnecessary medical resource consumption can be reduced by increasing the follow-up interval of pancreatic cyst patients with low risk of malignancy or not following them at all. To this end, in addition to imaging characteristics of pancreatic cysts, which are currently suggested as risk factors for malignancy in most guidelines for pancreatic cysts, differential diagnosis of pancreatic cysts based on new biomarkers such as genetic mutations and malignant risk assessment are necessary. Therefore, in this study, the investigators comprehensively analyze the blood, pancreatic cyst fluid, and pancreatic cyst tissue of patients with pancreatic cysts to explore biomarkers including genetic mutations that are helpful in the differential diagnosis of pancreatic cyst and the diagnosis of malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic cyst patients undergoing cyst aspiration or biopsy or surgical resection
* Patients who gave written informed consent

Exclusion Criteria:

* Anyone who has not signed a written consent form.
* Patients deemed unsuitable for research (severe infection, drug abuse, severe mental illness, etc.)

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Pancreatic cyst patients undergoing cyst aspiration or biopsy or surgical resection
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2028-05-15 (Estimated); Study Completion 2030-05-15 (Estimated)

PRIMARY OUTCOMES:
Genetic variants of pancreatic cysts associated with malignancy assessed by next-generation sequencing | Through study completion, an average of 3 years
  Genetic variants showing significant differences between pancreatic cysts with high-grade dysplasia or invasive cancer and the remaining pancreatic cysts, assessed through next-generation sequencing

SECONDARY OUTCOMES:
Genetic variants that differentiate mucinous from serous cysts assessed by next-generation sequencing | Through study completion, an average of 3 years
  Genetic variants indicating significant differences between mucinous and serous cysts, as evaluated through next-generation sequencing

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No